CLINICAL TRIAL: NCT07153445
Title: Phase II Clinical Trial of Chemotherapy + Atezolizumab for Stage IIIa and IIIb Non-small Cell Lung Cancer Followed by Atezolizumab as Adjuvant Treatment After Surgery and Atezolizumab as Maintenance Treatment for Non-resected Patients After Chemoradiotherapy
Brief Title: Neoadjuvant Treatment With Atezolizumab and Atezolizumab as Maintenance for the Treatment of Stage III Non Small-Cell Lung Cancer (NSCLC)
Acronym: ATHENEA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación GECP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GECP 23/02_ATHENEA; 2024-515984-68-00 (EU CTIS Number)
Record Dates: First submitted 2025-07-24; First posted 2025-09-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Non Small Cell Lung Cancer; Stage IIIA Lung Cancer; Stage IIIB Lung Cancer
Keywords: Non small cell lung cancer; Atezolizumab; Non-resected lung cancer; Adjuvant treatment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — atezolizumab; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: Neoadjuvant/Induction treatment (Experimental): Neoadjuvant/Induction treatment prior to surgery:
  * Atezolizumab
  * Paclitaxel:
  * Carboplatin
  After assessment by a multidisciplinary team who will decide on the best post-induction treatment
  Interventions: Drug: Atezolizumab; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Atezolizumab — Patients will receive atezolizumab administered by intravenous infusion in a monitored setting where there is immediate access to trained personnel and adequate equipment/medicine to manage potentially serious reactions.
  Other Names: Tecentriq
Drug: Paclitaxel — Neoadjuvant / induction treatment:
  Atezolizumab Paclitaxel Carboplatin
  Neoadjuvant / induction treatment 3 cycles will be administered prior to the assessment for surgery.
  Route of administration Paclitaxel: Intravenous infusion.
  Guidelines of Paclitaxel administration: Paclitaxel must be administered by infusion over 3 hours in dextrose (D5W) or normal saline (NS). The concentration must not exceed 1.2 mg/ml.
  Other Names: Taxol
Drug: Carboplatin — Neoadjuvant / induction treatment:
  Atezolizumab Paclitaxel Carboplatin*
  *Infusion according to the standard of each center
  Neoadjuvant / induction treatment 3 cycles will be administered prior to the assessment for surgery.
  Route of administration Carboplatin: Intravenous infusion. Guidelines of Carboplatin administration: According to the standard of each center.
  Other Names: Paraplatin

SUMMARY:
This is an open-label, phase II, multi-centre clinical trial. 97 Patients with stage IIIA and IIIB non-small cell lung cancer will be enrolled.

The treatment is Atezolizumab + Paclitaxel + Carboplatin 3 cycles as neoadjuvant/induction treatment. After the induction treatment every patient will be evaluated by a multidisciplinary team in each participant hospital to decide if the patient is candidate for surgery or not.

Depending on the decision each patient will be treated in a different way. The primary objective is to evaluate the Progression free survival (PFS). The total trial duration will be 10 years approximately. Patient accrual is expected to be completed within 2 years. Two years of treatment, 5 years of follow up, and 4-6 months of close-out.

DETAILED DESCRIPTION:
The study ATHENEA is a phase II clinical trial intending to enroll 97 patients, who will receive Atezolizumab + Paclitaxel + Carboplatin as induction/neoadjuvant treatment. After the induction treatment all patients will be evaluated by a multidisciplinary team in each participant hospital to decide if the patient is candidate for surgery or not.

Depending on the decision each patient will be treated in a different way.

The study is an open-label, phase II, multicenter clinical trial for previously untreated adult patients with stage to IIIA and IIIB non-small cell lung cancer.

The primary objective is to evaluate the Progression free survival (PFS) in the intent-to-treat population.

Progression free survival (PFS) defined as the time from initiation of treatment to the occurrence of disease progression or death.

The total trial duration will be 10 years approximately. Approval-start up: 4-6 months. Patient accrual is expected to be completed within 2 years. Two years of treatment, 5 years of follow up, and close-out: 4-6 months. The study will end once survival follow-up has concluded.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated patients with histologically- or cytologically- documented Non Small-Cell Lung Cancer (NSCLC) who present stage IIIA - IIIB disease (according to 8th version of the International Association for the Study of Lung Cancer Staging Manual in Thoracic Oncology)
* Confirm the absence of distant disease
* ECOG (Performance status) 0-1
* Adequate hematologic and organ function
* All patients are notified of the investigational nature of this study and signed a written in-formed consent in accordance with institutional and national guidelines, including the Declaration of Helsinki prior to any trial-related intervention
* Adequate lung function
* Patients aged > 18 years
* For female patients of childbearing potential, agreement (by patient and/or partner) to use a highly effective form(s) of contraception
* For male patients with female partners of childbearing potential, agreement (by patient and/or partner) to use a highly effective form of contraception
* Oral contraception should always be combined with an additional contraceptive method
* Women who are not postmenopausal or surgically sterile must have a negative serum pregnancy test result within 8 days prior to initiation of study drug.
* Patient capable of proper therapeutic compliance and accessible for correct follow-up

Exclusion Criteria:

* Patients mutation or an amplification in the EGFRgene, ALK fusion oncogene.
* Known STK-11 ligand alterations, MDM2 amplifications or ROS1 translocations.
* Weight loss >10% within the previous 3 months.
* Patients that receive previous treatment with antineoplasic drugs, chest radiotherapy, or previous surgery for lung cancer.
* Malignancies other than Non Small-Cell Lung Cancer (NSCLC) within 3 years prior to enrolment
* Pleural or pericardial effusion
* Known hypersensitivity or allergy to atezolizumab formulation.
* History of autoimmune disease or lung disease
* Positive test for human immunodeficiency viruses (HIV)
* Patients with active hepatitis B or hepatitis C or psitive for hepatitis C virus.
* Active tuberculosis.
* Symptomatic neuropathy grade > 1 according to Common Terminology Criteria for Adverse Events (CTCAE) v5.0
* Severe infections within 4 weeks prior to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2035-05-02 (Estimated); Study Completion 2035-05-02 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | From the date of randomization until end of follow up, up to 60 months.
  Progression free survival (PFS) defined as the time from initiation of treatment to the occurrence of disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.

SECONDARY OUTCOMES:
Resectability rate (%) | From the date of randomization until end of follow up, up to 60 months.
  Resectability rate defined as the percentage of patients resected divided by the total number of patients who received neoadjuvant treatment.
Pathological complete response (pCR) | From the date of randomization until end of surgery, up to 6 months
  Pathological complete response (pCR) is defined as the absence of residual viable tumor on hematoxylin and eosin evaluation of the complete resected specimen
Overall survival (OS) | From the date of randomization until end of follow up, up to 60 months.
  Overall survival (OS) defined as the time which begins at the start of treatment and up to the time of death or last follow up

CONTACTS AND LOCATIONS:
Overall Officials: Mariano Provencio, MD, Study Chair — President of Grupo Español de Cáncer de Pulmón
Locations (21):
- Spain (21):
  - Hospital General Universitario Dr. Balmis de Alicante, Alicante, Alicante
  - ICO Badalona, Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d' Hebron, Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Barcelona
  - Hospital Parc Taulí, Barcelona, Barcelona
  - Hospital De Basurto, Bilbao, Bilbao
  - Hospital Univ. De Jerez De La Frontera, Jerez de la Frontera, Cadiz
  - ICO Girona, Hospital Josep Trueta, Girona, Girona
  - Hospital Universitario Clinico San Cecilio, Granada, Granada
  - Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Hospital Universitari de Gran Canària Doctor Negrín, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Lucus Augusti, Lugo, Lugo
  - Hospital Universitario Fundación Jiménez Díaz, Madrid, Madrid
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Universitari Son Llatzer, Palma de Mallorca, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona, Pamplona
  - Hospital Universitario Salamanca, Salamanca, Salamanca
  - Hospital Universitario Nuestra Señora La Candelaria, Santa Cruz de Tenerife, Santa Cruz de Tenerife
  - Hospital Universitario Virgen Del Rocio, Seville, Sevilla
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital General Universitario de Valencia, Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Description Web page of the sponsor where users can find more information about Fundación GECP studies — http://www.gecp.org